CLINICAL TRIAL: NCT01253460
Title: A Phase II Clinical Trial of Sapacitabine, Cyclophosphamide, and Rituximab (SCR) for Relapsed Patients With Chronic Lymphocytic Leukemia / Small Lymphocytic Lymphoma (CLL/SLL) and Deletion 11q22-23 by FISH
Brief Title: Sapacitabine, Cyclophosphamide, Rituximab for Relapsed Chronic Lymphocytic Leukemia, Small Lymphocytic Lymphoma (CLL/SLL) With Deletion (11q22-23)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Accrual not met
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cyclacel Pharmaceuticals, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0516; NCI-2011-00119 (Registry Identifier: NCI CTRP); 5P01CA081534 (NIH)
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Leukemia
Keywords: Chronic Lymphocytic Leukemia; CLL; Small Lymphocytic Lymphoma; SLL; Cyclophosphamide; Rituximab; Sapacitabine; Cytoxan; Neosar; Rituxan
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclophosphamide; Rituximab; sapacitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cyclophosphamide, Rituximab + Sapacitabine (Experimental): After Sapacitabine 350 mg orally Days 1-3, Cyclophosphamide 250 mg/m2 IV 2 hours, followed by Rituximab 375 mg/m2 IV Day 3, Course 1, and 500 mg/m2 Day 1, subsequent courses.
  Interventions: Drug: Cyclophosphamide; Drug: Rituximab; Drug: Sapacitabine

INTERVENTIONS:
Drug: Cyclophosphamide — 250 mg/m2 by vein (IV) over 30 minutes, 2 hours following the dose of Sapacitabine on days 1, 2, and 3 of each 28 day course.
  Other Names: Cytoxan; Neosar
Drug: Rituximab — 375 mg/m2 by vein over 6 - 8 hours on day 3 of course 1 after cyclophosphamide, then at 500 mg/m2 on day 1, after cyclophosphamide for subsequent courses. Each course is 28 days.
  Other Names: Rituxan
Drug: Sapacitabine — 350 mg flat dose by mouth in the morning of days 1,2, and 3 of each 28 day course.

SUMMARY:
The goal of this clinical research study is to learn if sapacitabine given in combination with 2 standard drugs (cyclophosphamide and rituximab) can help to control CLL and SLL. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Sapacitabine and cyclophosphamide are designed to damage the DNA (genetic material) of cancer cells, which may cause the cancer cells to die.

Rituximab is designed to attach to cancer cells and damage them, which may cause the cancer cells to die. It is also designed to cause the immune system to attack cancer cells.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive sapacitabine by mouth 1 time a day on Days 1-3 of each 28-day cycle. Try to take sapacitabine at least 1 hour before or 2 hours after a meal. On Days 1-3 of each cycle, you will also receive cyclophosphamide by vein over 30 minutes, starting 2 hours after you take sapacitabine.

On Day 3 of Cycle 1 and Day 1 of Cycles 2 and beyond, you will receive rituximab by vein over 6-8 hours.

If side effects occur, the study doctor may decide to lower your study drug doses. If you have side effects during a dose, the study staff will check you for any other problems for 2 hours after the dose.

Other Drugs:

On Days 1-14 of Cycle 1, you will take allopurinol by mouth 1 time a day to lower the risk of kidney damage.

Before each dose of cyclophosphamide, you will receive Zofran (ondansetron) by vein over a few seconds to lower the risk of nausea.

About 30-60 minutes before each dose of rituximab, you will take Tylenol (acetaminophen) and Benadryl (diphenhydramine hydrochloride) by mouth to lower the risk of side effects such as fever and chills.

Study Visits:

On Day 1 of each cycle:

* Blood (about 1-2 tablespoons) will be drawn for routine tests.
* You will also have a physical exam, including measurement of your vital signs, except Cycle 1.
* You will be asked about any side effects you may have had.

On Days 8 and 22 of Cycle 1, and on Day 15 of every cycle:

* Blood (about 1-2 tablespoons) will be drawn for routine tests.
* You will be asked about any side effects you may have had.

If your disease has had a good response and the doctor thinks it is needed to check the status of the disease, you will have a bone marrow aspiration and biopsy and a CT scan of the chest, abdomen and pelvis prior to Cycle 4 and possibly every other cycle after that (Cycles 6, 8, 10, and so on).

Length of Study:

Once your doctor thinks the disease has had its best response, you may receive 2 more cycles of study therapy after that. You will no longer be able to receive the study drugs if the disease gets worse or intolerable side effects occur.

End-of-Treatment Visit:

The following tests and procedures will be performed after your last cycle of study drugs:

* You will have a physical exam, including measurement of your vital signs.
* Blood (about 2 tablespoons) will be drawn for routine tests.

Follow-Up Visits:

At 2 and 6 months and 1 and 2 years after your last dose of study drugs:

* You will be asked about any side effects you may have had and any drugs you may be taking.
* You will have a physical exam, including measurement of your vital signs.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* If the doctor thinks the disease has completely responded, you will have a CT scan of the neck, chest, abdomen, and pelvis to confirm the response. You will also have a bone marrow aspiration and biopsy to confirm the response.

At 3 years after your last dose of study drugs and 1 time a year from then on:

* You will be asked about any side effects you may have had and any drugs you may be taking.
* You will have a physical exam, including measurement of your vital signs.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* You will have a bone marrow aspiration and biopsy if the doctor decides it is needed to check the status of the disease.

If the doctor thinks it is needed anytime during follow-up, you will have a CT scan of the neck, chest, abdomen, and pelvis to check the status of the disease.

Starting at Year 3, the follow-up tests and procedures can be done by your local doctor if that is more convenient to you. The test results should be sent to MD Anderson.

You should tell your study doctor or staff if you start another cancer treatment during follow-up. If that occurs, your follow-up in this study will stop.

This is an investigational study. Sapacitabine is not FDA approved or commercially available. It is currently being used for research purposes only. Cyclophosphamide and rituximab are FDA approved and commercially available to treat CLL and SLL. The combination of sapacitabine, cyclophosphamide, and rituximab is investigational.

Up to 40 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a diagnosis of CLL/SLL and be previously treated
2. Patients must have had Fluorescence in situ Hybridization (FISH) evaluation of leukemia cells within 3 months without intervening treatment demonstrating deletion 11q22-23
3. Patients must have an indication for treatment by 2008 International Workshop on Chronic Lymphocytic Leukemia (IWCLL) Criteria
4. Age >/= 18 years
5. Eastern Cooperative Oncology Group (ECOG)/Zubrod performance status </= 2
6. Adequate renal and hepatic function as indicated by all the following: serum creatinine </= 2 mg/dL AND; alanine aminotransferase (ALT) </= 2.5 times upper limit of normal; AND total bilirubin </= 2.5 times upper limit of normal
7. Patients must have an Absolute neutrophil count (ANC) >/= 500/uL, Hemoglobin (HGB) >/= 8 gm/dL, Platelets (PLT) count >/= 20K/uL, unless attributed to marrow infiltration with CLL
8. Patients must give written informed consent
9. Patients of childbearing potential (females who have not been postmenopausal for at least 12 consecutive months or who have not undergone previous surgical sterilization or males who have not been surgically sterilized) must be willing to practice birth control during the study

Exclusion Criteria:

1. Pregnant or breast-feeding females
2. Significant co-morbidity indicated by major organ system dysfunction
3. Active infection, uncontrolled with intravenous antibiotics
4. Uncontrolled autoimmune hemolytic anemia (AIHA) or immune thrombocytopenia purpura (ITP)
5. Treatment including chemotherapy, chemoimmunotherapy, monoclonal antibody therapy, radiotherapy, high-dose corticosteroid therapy (prednisone >/= 60 mg daily, or equivalent), or immunotherapy within 3 weeks prior to enrollment or concurrent with this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-08-22 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2019-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G. Wierda, MD, PHD, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 8/22/2011 to 12/19/2013
Period: Overall Study
Arm/Group | Cyclophosphamide, Rituximab + Sapacitabine
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cyclophosphamide, Rituximab + Sapacitabine
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Patients evaluated for response by 2008 International Workshop on Chronic Lymphocytic Leukemia [IWCLL] overall response criteria before course 4, then after every 2 courses, and at end of treatment (2 months after last course). Overall Response Rate (ORR) = Complete Response (CR) + Partial Response (PR). Complete response is the absence of signs and symptoms, normalization of peripheral blood and bone marrow and lymph nodes 1.5 cm in diameter or smaller on CT scan. Partial response is at least 50% reduction in disease signs and symptoms, a 50% improvement in peripheral blood and greater than or equal to 50% reduction in lymph nodes.
Time Frame: 84 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide, Rituximab + Sapacitabine
Number analyzed (Participants) | 18
Participants | 8

2. Secondary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Up to 8.5 years
Measure: Median (Full Range); unit: Months
Arm/Group | Cyclophosphamide, Rituximab + Sapacitabine
Number analyzed (Participants) | 18
Months | 31 [2 to 92]

ADVERSE EVENTS:
Time Frame: Up to 8.5 years
Arm/Group | Cyclophosphamide, Rituximab + Sapacitabine
All-Cause Mortality (participants affected / at risk) | 2/18
Serious Adverse Events (participants affected / at risk) | 7/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide, Rituximab + Sapacitabine (N=18)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Neutropenic Fever (Infections and infestations) | 1 (1)
Dyspena (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Leukemia Secondary to Chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Renal Calculi (Renal and urinary disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Neoplasms benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Soft Tissue Infection (Infections and infestations) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lymph node pain (General disorders) | 1 (1)
Sycnope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide, Rituximab + Sapacitabine (N=18)
Abdominal Distension (Gastrointestinal disorders) | 3 (3)
Anorexia (Gastrointestinal disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 4 (17)
Neutropenia (Blood and lymphatic system disorders) | 12 (48)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (33)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chills (General disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 3 (3)
Dehydration (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Dizziness (Nervous system disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Edema, Limbs (Blood and lymphatic system disorders) | 4 (4)
Epistaxis (Blood and lymphatic system disorders) | 3 (3)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 4 (4)
Headache (General disorders) | 2 (2)
Hot Flashes (Endocrine disorders) | 5 (5)
Infusion Reaction (Investigations) | 2 (2)
Infection (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (7)
Pain, arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain, Extremity (General disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Elevated Creatinine (Metabolism and nutrition disorders) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (3)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-06-28): https://cdn.clinicaltrials.gov/large-docs/60/NCT01253460/Prot_SAP_000.pdf